CLINICAL TRIAL: NCT04161339
Title: Effect of Hydroxychloroquine on Endothelial Function: a Clinical Trial
Brief Title: Anti-Inflammatory Drug and Endothelial Function
Acronym: HOLD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Collaborators: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5351/17
Record Dates: First submitted 2019-10-29; First posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: Cardiovascular Diseases; Endothelial Dysfunction; Sleep Apnea; Atherosclerosis; Coronary Artery Disease
MeSH Terms: conditions — Cardiovascular Diseases; Sleep Apnea Syndromes; Atherosclerosis; Coronary Artery Disease | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxychloroquine (Experimental): 400mg/daily of hydroxychloroquine for 8 weeks
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Hydroxychloroquine — 400mg/daily of hydroxychloroquine for 8 weeks
  Arms: Hydroxychloroquine
Drug: Placebo oral tablet — Amido pills/daily for 8 weeks
  Arms: Placebo

SUMMARY:
In this randomized double-blinded clinical trial, 400mg of hydroxychloroquine will be given daily to people over the age of 65 years with moderate-severe obstructive sleep apnea for 8 weeks. The aim of this study is to test whether hydroxychloroquine can improve endothelial function.

DETAILED DESCRIPTION:
Sleep apnea and coronary artery disease are prevalent and relevant diseases due to their morbidity and mortality. The mechanism by which sleep apnea leads to coronary artery disease remains unclear. It is known that intermittent hypoxia, the main characteristic of sleep apnea, leads to inflammation and consequently may lead to endothelial dysfunction. Endothelial dysfunction precedes the development of atherosclerotic disease and the occurrence of cardiovascular events. Agents that potentially act to improve endothelial function may assist in the prevention of cardiovascular events. Patients using immunomodulators due to rheumatic diseases have a lower prevalence of cardiovascular diseases. However, the cardioprotective effect of these drugs in patients without autoimmune diseases is not known. Hydroxychloroquine (HCQ) is an immunomodulator used in the treatment of rheumatoid arthritis and systemic lupus erythematosus. In addition to its anti-inflammatory properties, HCQ reduces cholesterol and glycemia levels and has antithrombotic effects. The drug is inexpensive and widely available. The adverse effects of HCQ are rare and occur more frequently when using high doses.

ELIGIBILITY:
Inclusion Criteria:

* Apnea-Hypopnea index of 15 events/hour or higher

Exclusion Criteria:

* Contraindication for hydroxychloroquine (retinopathy, chronic liver disease, chronic renal disease)
* Rheumatologic disease

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in endothelial function measured by peripheral artery tonometry in the reactive-hyperemia index (RHI) scale | before and after eight weeks of treatment with hydroxychloroquine
  The reactive-hyperemia index (RHI) scale ranges from -0.4 to 1.6. Below -0.51 being endothelial dysfunction, a higher score indicates a better endothelial function
Change in endothelial function measured by flow-mediated dilation (%FMD-response) | before and after eight weeks of treatment with hydroxychloroquine
  The FMD-response will be calculated as the variation in post-hyperaemia brachial artery diameter from baseline, measured in relative (percentage) change. A mean improvement in flow mediated dilatation of at least 2% would usually be required to detect a treatment benefit.

SECONDARY OUTCOMES:
Change in fasting glucose blood levels (mg/dL) | before and after eight weeks of treatment with hydroxychloroquine
Change in glycosylated hemoglobin blood levels (%) | before and after eight weeks of treatment with hydroxychloroquine
Change in Lipidic profile | before and after eight weeks of treatment with hydroxychloroquine
  Determined by total cholesterol, HDL-cholesterol and triglycerides blood levels (mg/dL)
Change in C-reactive protein (CRP) blood levels (mg/L) | before and after eight weeks of treatment with hydroxychloroquine
  The risk of developing cardiovascular disease is quantified as follows:
  low: CRP level under 1.0 mg/L average: between 1.0 and 3.0 mg/L high: above 3.0 mg/L
Change in neutrophils lymphocytes ratio (NLR) | before and after eight weeks of treatment with hydroxychloroquine
  calculated by dividing the number of neutrophils by number of lymphocytes. The mean range of healthy adult subjects is between 0.78 and 3.53.
Change in Autonomic Nervous System | before and after eight weeks of treatment with hydroxychloroquine
  The data will be collected through the system of acquisition of pressure waves in a continuous and non-invasive way by the Finometer® system, through a cuffing installed in the middle finger, taking this signal to an analog-to-digital signal converter. The pulse pressure signal will be acquired at 1000 Hz, continuously and non-invasively, supine (10 minutes) in a quiet environment, with controlled temperature (± 23 ° C) and illumination. The collected data will be saved in the software BeatsScope® and LabChart®, from which will be extracted the systograms for analysis.
Change in apnea/hypopnea index | before and after eight weeks of treatment with hydroxychloroquine
  Apnea/Hypopnea index is provided by home respiratory polygraphy, ranging from 0-highest events/hour, zero-5 eventos/hour being normal and above 5 events/hour being abnormal

CONTACTS AND LOCATIONS:
Overall Officials: Denis Martinez, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tedesco Silva LM, Cortes A, Rossi B, Boll L, Waclawovsky G, Eibel B, Cadaval Goncalves S, Irigoyen MC, Martinez D. Effects of Hydroxychloroquine on endOthelial function in eLDerly with sleep apnea (HOLD): study protocol for a randomized clinical trial. Trials. 2021 Sep 17;22(1):638. doi: 10.1186/s13063-021-05610-0. PMID 34535165